CLINICAL TRIAL: NCT05052593
Title: Effects of Compressive Myofascial Release of Vastus Lateralis on Lateral Patellar Tracking in Patients With Knee Osteoarthritis.
Brief Title: Compressive Myofascial Release in Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/00870 Rubia Batool
Record Dates: First submitted 2021-06-11; First posted 2021-09-22 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2021-09

CONDITIONS: Osteoarthritis, Knee
Keywords: knee osteoarthritis; compressive myofascial release; lateral patellar tracking
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: the purpose of this study is to compare the effects of compressive myofascial release on lateral patellar tracking inpatients with knee osteoarthritis. an RCT trial was conducted at Railway general hospital, Ahad medi care clinics and physiotherapy centre rawat and THP Bahria town phase 6.sample size was 52 calculated through open-epi tool. participants divided into control and experimental group.participants diagnosed with grade 2and 3 K&L classification of knee OA included.
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Compressive myofascial release (Experimental): . patients in this group will receive treatment through CMR that includes shaking the muscle belly of vastus lateralis for 30 seconds. Then the hip is fully extended on treatment table and CMR is applied on Vastus lateralis muscle for 1 minute. Treatment consists of broad strokes applied with clinicians knuckles to release superficial restrictions, followed by more specific strokes applied with clinicians' thumb on tight muscle. Strokes are applied at a contact point of 45 degree. with pressure directed from distal to proximal.
  Conventional treatment of Hot pack and Tens for 20 minutes, Range of motion exercises (knee flexion and extension ROM's), Stretching exercises (3sets, 10 reps for 5 second hold)
  Interventions: Other: compressive myofascial release
- Conventional treatment (Active Comparator): Patients in this group will receive treatment of Hot pack and Tens for 20 minutes, Range of motion exercises (knee flexion and extension ROM's), Stretching exercises (3sets, 10 reps for 5 second hold)
  Interventions: Other: conventional treatment group

INTERVENTIONS:
Other: compressive myofascial release — Patients in this group will receive treatment through CMR that includes shaking the muscle belly of vastus lateralis for 30 seconds. Then the hip is fully extended on treatment table and CMR is applied on Vastus lateralis muscle for 1 minute. Treatment consists of broad strokes applied with clinicians knuckles to release superficial restrictions, followed by more specific strokes applied with clinicians' thumb on tight muscle. Strokes are applied at a contact point of 45 degree. With pressure directed from distal to proximal.
  Arms: Compressive myofascial release
Other: conventional treatment group — Patients in this group will receive treatment of Hot pack and Tens for 20 minutes, Range of motion exercises (knee flexion and extension ROM's), Stretching exercises (3sets, 10 reps for 5 second hold)
  Arms: Conventional treatment

SUMMARY:
The purpose of the study is to compare the effects of compressive myofascial release and conventional knee osteoarthritis treatment to correct lateral patellar tracking. A randomized control trial was conducted at Railway General Hospital, Ahad Medicare clinics and physiotherapy Centre and The Health Professional physiotherapy clinic Bahria town phase 6. The sample size was 52 calculated through open-epi tool. The participants were divided into two interventional groups each having 26 participants. The study duration was six months. Sampling technique applied was non probability convenient sampling for recruitment and group randomization using sealed enveloped method. Only participants who were 50 years above with grade 2 and 3 knee osteoarthritis were included in the study. Tools used in this study are Q angle, numeric pain rating scale, goniometry and WOMAC questionnaire, Self structured Questionnaire. Data was collected at baseline, at the end of 3rd session and 6th session. Data analyzed through SPSS version 23.

DETAILED DESCRIPTION:
knee osteoarthritis is commonly manifested as decreased joint space, sub chondral bone sclerosis, bony spur formation, cartilage loss and mainly lateral patellar tracking(2).Lateral patellar tracking is a condition in which patellar move laterally in relation to femoral groove on flexion and extension(4). Patellofemoral disorders are very common in patients of knee OA. One of the very common manifestation of which is lateral patellar tracking(5). Patella move laterally due to certain disorders of knee that include patellofemoral pain syndrome and anterior knee pain. Q-angle is used as an indicator of patellofemoral pain syndrome. When Q angle exceeds its normal limit i.e. 15-20 degrees it leads to lateral mal positioning of patella(6). Rozenfeld, E et al. in 2019 conducted a cross sectional study with a diagnosis of anterior knee pain that suggests highest prevalence of myofascial trigger points in distal vastus lateralis and mid and distal vastus lateralis. It also reported that presence of trigger points in anterior knee pain(7). There are several techniques that are used to release trigger points.

ELIGIBILITY:
Inclusion Criteria:

* Includes diagnosed cases of knee osteoarthritis
* Grades 2-3 according to the Kellgren and Lawrence method of grading(1)
* Includes patients from the age group of 50 years and above(3)
* Includes knee osteoarthritis patients with lateral tracking of patella which will assessed through Q angle test(4)

Exclusion Criteria:

* history of recent trauma to knee
* History of hip disease
* Past history of knee surgery/arthroplasty
* Intraarticular corticosteroid injection

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2020-08-14 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Western Ontario and McMaster Universities Arthrosis Index (WOMAC) scale: | 4th Week
  Western Ontario and McMaster Universities Arthrosis Index WOMAC was first developed in 1988 by Bellamy for use in patients with hip and knee osteoarthritis is a self-administered tool comprising of 24 items divided into 3 sub scales. It was used to assess pain, stiffness and physical function in knee osteoarthritis patients which were allocated in the study. Patient's pain is assessed by asking about intensity of pain in different positions including pain intensity at rest through 5 questions. Patient is asked about stiffness level in the morning and evening (2 questions). Patients is also assessed for difficulty doing several daily and self-care activities in 17 different questions. Each item in sub scale carries maximum score of 4 and minimum score of 0. Overall score of WOMAC scale is 100 with a cutoff value of 39. In first session, 2 and 4 weeks after treatment sessions.

SECONDARY OUTCOMES:
Numeric Pain Rating Scale: | 4th Week
  Numeric pain rating scale is a type of scale which is used to measure pain intensity. It is easy to use as the patient can report the intensity of his/her pain by simply looking at the scale. The scale has ratings from 0 to 10, where the point 0 means no pain, the points 1, 2 and 3 measure pain of mild intensity, the points 4,5 and 6 measure pain of moderate intensity and the demarcations 7,8,9 and 10 measures severe intensity of pain. It was used in this study to measure the intensity of knee joint pain reported by each patient. Numeric pain rating scale is preferred over visual analog scale for use in elderly individuals. The patients are asked about the subjective examination of intensity of pain after describing the demarcations present on the scale to the patient about the maximum and minimum values. In first session, 2 and 4 weeks after treatment sessions.

OTHER OUTCOMES:
Functional Reach Test: | 4th Week
  Functional reach test was utilized to determine instability present in the patient, in particular, dynamic standing balance was measured. During this test the participant was advised to stand next to the wall, not leaning against the wall, feet were at a comfortable distance apart. Care must be taken to assess the patient who is elderly and the one who has balance issues. Continuous supervision throughout the test is necessary and therapist must be there to help patient achieve and maintain the position. The participant was asked to flex the dominant arm to 90 degree and reach as much forward as possible without overbalancing. In first session, 2 and 4 weeks after treatment sessions.
Measurement Quadriceps Angle: | 4th Week
  Q-angle measurement was used to assess lateral patellar tilting that is the primary objective. Q angle measurement with a goniometer is a standardized protocol and test-retest reliability was found out through intra-tester reliability study which included 52 adults with no history of knee injury. Reliability came out to be to be 0.88(45). Q-angle at knee is assessed by asking the patient to assume supine position with hip and knee extended at treatment table, arms by the side of the body, foot is always in neutral position with isometric contraction of rectus femoris. The bony landmarks that are used to assess Q-angle are anterior superior iliac spine, tibial tuberosity, and patella. In first session, 2 and 4 weeks after treatment sessions.
Goniometry: | 4th Week
  It was used to assess knee joint range of motion with a reliable and valid tool goniometer. It has a fulcrum and 2 arm that are used to measure the angle. Reliability is found out to be 0.92-0.99 which is categorized as good reliability.
  In this study goniometer was used to find out Q-angle, knee flexion ROM and knee extension ROM for each patient in both control and experimental groups. For Q-angle measurement the center point was placed at center of patella, the proximal arm was placed parallel to anterior superior iliac spine and distal arm was placed at tibial tuberosity of the patient. In first session, 2 and 4 weeks after treatment sessions.

CONTACTS AND LOCATIONS:
Overall Officials: Lal Gul Khan, MScPT, Principal Investigator — Riphah International University
Locations (2):
- Pakistan (2):
  - Bone and joints centre, Rawalpindi, Punjab Province
  - Railway General Hospital, Rawalpindi, Punjab Province

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brandt KD, Fife RS, Braunstein EM, Katz B. Radiographic grading of the severity of knee osteoarthritis: relation of the Kellgren and Lawrence grade to a grade based on joint space narrowing, and correlation with arthroscopic evidence of articular cartilage degeneration. Arthritis Rheum. 1991 Nov;34(11):1381-6. doi: 10.1002/art.1780341106. PMID 1953815
- [Background] Zhang Y, Jordan JM. Epidemiology of osteoarthritis. Clin Geriatr Med. 2010 Aug;26(3):355-69. doi: 10.1016/j.cger.2010.03.001. PMID 20699159
- [Background] Hunter DJ, Felson DT. Clinical review: osteoarthritis. British Medical Journal [periódico online]. 2006:639-42.
- [Background] Doucette SA, Goble EM. The effect of exercise on patellar tracking in lateral patellar compression syndrome. Am J Sports Med. 1992 Jul-Aug;20(4):434-40. doi: 10.1177/036354659202000412. PMID 1415887
- [Background] Ntagiopoulos PG, Dejour D. Patellofemoral Pain, Instability, and Arthritis. Patellofemoral Pain, Instability, and Arthritis: Clinical Presentation, Imaging, and Treatment. 2020:1.
- [Background] Turkmen F, Acar MA, Kacira BK, Korucu IH, Erkocak OF, Yolcu B, Toker S. A new diagnostic parameter for patellofemoral pain. Int J Clin Exp Med. 2015 Jul 15;8(7):11563-6. eCollection 2015. PMID 26379982
- [Background] Rozenfeld E, Finestone AS, Moran U, Damri E, Kalichman L. The prevalence of myofascial trigger points in hip and thigh areas in anterior knee pain patients. J Bodyw Mov Ther. 2020 Jan;24(1):31-38. doi: 10.1016/j.jbmt.2019.05.010. Epub 2019 May 14. PMID 31987560
- [Background] Stanek J, Sullivan T, Davis S. Comparison of Compressive Myofascial Release and the Graston Technique for Improving Ankle-Dorsiflexion Range of Motion. J Athl Train. 2018 Feb;53(2):160-167. doi: 10.4085/1062-6050-386-16. Epub 2018 Jan 26. PMID 29373060
- [Background] Vijayakumar M, Jaideep A, Khankal R. Effectiveness of Compressive Myofascial Release Vs Instrument Assisted Soft Tissue Mobilization in Subjects with Active Trigger Points of the Calf Muscle Limiting Ankle Dorsiflexion. International Journal of Health Sciences and Research. 2019;9(4):98-106
- [Background] De Souza IG, Pavan Kumar G. Effect of Releasing Myofascial Chain in Patients with Patellofemoral Pain Syndrome-A Randomized Clinical Trial. Int J Cur Res Rev| Vol. 2020;12(08):5.
- [Background] Kohn MD, Sassoon AA, Fernando ND. Classifications in Brief: Kellgren-Lawrence Classification of Osteoarthritis. Clin Orthop Relat Res. 2016 Aug;474(8):1886-93. doi: 10.1007/s11999-016-4732-4. Epub 2016 Feb 12. No abstract available. PMID 26872913
- [Background] Ferre IM, Roof MA, Anoushiravani AA, Wasterlain AS, Lajam CM. Understanding the Observed Sex Discrepancy in the Prevalence of Osteoarthritis. JBJS Rev. 2019 Sep;7(9):e8. doi: 10.2106/JBJS.RVW.18.00182. No abstract available. PMID 31567717
- [Background] Nguyen TV. Osteoarthritis in southeast Asia. International Journal of Clinical Rheumatology. 2014.
- [Background] Jordan JM, Helmick CG, Renner JB, Luta G, Dragomir AD, Woodard J, Fang F, Schwartz TA, Abbate LM, Callahan LF, Kalsbeek WD, Hochberg MC. Prevalence of knee symptoms and radiographic and symptomatic knee osteoarthritis in African Americans and Caucasians: the Johnston County Osteoarthritis Project. J Rheumatol. 2007 Jan;34(1):172-80. PMID 17216685
- [Background] Dor A, Kalichman L. A myofascial component of pain in knee osteoarthritis. J Bodyw Mov Ther. 2017 Jul;21(3):642-647. doi: 10.1016/j.jbmt.2017.03.025. Epub 2017 Apr 6. PMID 28750978
- [Background] Weiss L, DeForest B, Hammond K, Schilling B, Ferreira L. Reliability of goniometry-based Q-angle. PM R. 2013 Sep;5(9):763-8. doi: 10.1016/j.pmrj.2013.03.023. Epub 2013 Mar 22. PMID 23528815
- [Background] Alghadir AH, Anwer S, Iqbal A, Iqbal ZA. Test-retest reliability, validity, and minimum detectable change of visual analog, numerical rating, and verbal rating scales for measurement of osteoarthritic knee pain. J Pain Res. 2018 Apr 26;11:851-856. doi: 10.2147/JPR.S158847. eCollection 2018. PMID 29731662
- [Background] Shamsi M, Mirzaei M, Khabiri SS. Universal goniometer and electro-goniometer intra-examiner reliability in measuring the knee range of motion during active knee extension test in patients with chronic low back pain with short hamstring muscle. BMC Sports Sci Med Rehabil. 2019 Mar 22;11:4. doi: 10.1186/s13102-019-0116-x. eCollection 2019. PMID 30949343
- [Background] Lage PTS, Machado LAC, Barreto SM, de Figueiredo RC, Telles RW. Measurement properties of Portuguese-Brazil Western Ontario and McMaster Universities osteoarthritis index (WOMAC) for the assessment of knee complaints in Brazilian adults: ELSA-Brasil Musculoskeletal cohort. Rheumatol Int. 2020 Feb;40(2):233-242. doi: 10.1007/s00296-019-04496-1. Epub 2019 Dec 19. PMID 31858210
- [Background] Williams SB, Brand CA, Hill KD, Hunt SB, Moran H. Feasibility and outcomes of a home-based exercise program on improving balance and gait stability in women with lower-limb osteoarthritis or rheumatoid arthritis: a pilot study. Arch Phys Med Rehabil. 2010 Jan;91(1):106-14. doi: 10.1016/j.apmr.2009.08.150. PMID 20103404
- [Background] Duncan PW, Weiner DK, Chandler J, Studenski S. Functional reach: a new clinical measure of balance. J Gerontol. 1990 Nov;45(6):M192-7. doi: 10.1093/geronj/45.6.m192. PMID 2229941
- [Background] Hill KD, Bernhardt J, McGann AM, Maltese D, Berkovits D. A new test of dynamic standing balance for stroke patients: reliability, validity and comparison with healthy elderly. Physiotherapy Canada. 1996;48(4):257-62.
- [Background] Manheim CJ. The Myofascial Release Manual: SLACK; 2008
- [Background] Bennell KL, Ahamed Y, Bryant C, Jull G, Hunt MA, Kenardy J, Forbes A, Harris A, Nicholas M, Metcalf B, Egerton T, Keefe FJ. A physiotherapist-delivered integrated exercise and pain coping skills training intervention for individuals with knee osteoarthritis: a randomised controlled trial protocol. BMC Musculoskelet Disord. 2012 Jul 24;13:129. doi: 10.1186/1471-2474-13-129. PMID 22828288